CLINICAL TRIAL: NCT04781179
Title: Randomized, Controlled Study of the Effectiveness of Mental Contrasting and Implementation Intention in the Management of Apathy in Schizophrenia
Brief Title: Study of the Effectiveness of Mental Contrasting and Implementation Intention in the Management of Apathy in Schizophrenia
Acronym: COMEIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RECHMPL20_0447
Record Dates: First submitted 2021-02-19; First posted 2021-03-04 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2021-05

CONDITIONS: Schizophrenia; Apathy
Keywords: implementation intention; mental contrasting; apathy; schizophrenia; motivation
MeSH Terms: conditions — Schizophrenia; Lethargy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CM-II Technique (Experimental)
  Interventions: Behavioral: CM-II
- Psychoeducation (Placebo Comparator)
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: CM-II — It is an intervention of 4 two-hour sessions with a psychologist, MC-II technique
  Arms: CM-II Technique
Behavioral: Psychoeducation — It is an intervention of 4 two-hour sessions with a psychologist, psychoeducation
  Arms: Psychoeducation

SUMMARY:
Schizophrenia is a mental pathology that concerns 1% of the French population, characterized by heterogeneity of symptoms. One of them, apathy is defined as a multidimensional psychopathological state manifested by a decrease in motivation. This deficit is most common in schizophrenia and impacts the functional outcome of patients. To date, no treatment has shown a significant effect on this symptom. In other pathologies with a motivational deficit, the technique of Mental Contrasting and Implementation Intention (CM-II) showed interesting effects in improving motivation, reducing the effort related to the action.

The investigators aim to propose the CM-II technique to individuals with schizophrenia to improve apathy.

The investigators expected that the CM-II technique will allow an improvement of apathy which will have beneficial effects on other psychological factors (e.g., depressive symptoms). In addition, the implementation of the CM-II will provide help to global management.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and < 60 years old
* Diagnosis of schizophrenia according to DSM 5 criteria.
* Score greater than or equal to -18 on the Lille Apathy Rating Scale
* Ability to understand and speak French.
* Obligation to belong to or be a beneficiary of a social security scheme.
* Signature of the consent. If the participant has a representative, signature by the representative.

Exclusion Criteria:

* History of head injuries or neurological pathologies.
* Current treatment with sismotherapy or repetitive Transcranial Magnetic Stimulation (rTMS).
* Treatment targeted at and/or influencing negative symptoms (CBT, cognitive remediation), or therapeutic trial.
* Participant under safeguard of justice.
* Pregnant or breastfeeding woman.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-02-22 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Change of at least one class at the Lille Apathy Rating Scale (LARS) at 3 months | Change between Baseline and 3 months
  LARS (Sockeel et al. 2006, translated and validated in French by Yazbek et al. 2014) is a questionnaire semi-structured based on a multidimensional approach to apathy. It is composed of 33 grouped items in nine dimensions: activities of daily living, interests, taking initiative, interest in novelty, voluntary efforts, the intensity of emotions, worry, social life, and self-critical capability. Each item can be rated at 1 (no) or -1 (yes), a score of 0 is possible. if the answer is not classifiable. The total score on this scale ranges from -36 to +36 and allows for different classes: non-apathetic (score -36 to -22); tendency to apathy (-21 to -17); moderate apathy (-16 to -10); and severe apathy (-9 to +36).

SECONDARY OUTCOMES:
the improvement of at least one class at the Lille Apathy Rating Scale (LARS) at 1 month | Change between Baseline and 1 month
  LARS (Sockeel et al. 2006, translated and validated in French by Yazbek et al. 2014) is a questionnaire semi-structured based on a multidimensional approach to apathy. It is composed of 33 grouped items in nine dimensions: activities of daily living, interests, taking initiative, interest in novelty, voluntary efforts, the intensity of emotions, worry, social life, and self-critical capability. Each item can be rated at 1 (no) or -1 (yes), a score of 0 is possible. if the answer is not classifiable. The total score on this scale ranges from -36 to +36 and allows for different classes: non-apathetic (score -36 to -22); tendency to apathy (-21 to -17); moderate apathy (-16 to -10); and severe apathy (-9 to +36).
the improvement of at least one class at the Lille Apathy Rating Scale (LARS) at 6 months | Change between Baseline and 6 months
  LARS (Sockeel et al. 2006, translated and validated in French by Yazbek et al. 2014) is a questionnaire semi-structured based on a multidimensional approach to apathy. It is composed of 33 grouped items in nine dimensions: activities of daily living, interests, taking initiative, interest in novelty, voluntary efforts, the intensity of emotions, worry, social life, and self-critical capability. Each item can be rated at 1 (no) or -1 (yes), a score of 0 is possible. if the answer is not classifiable. The total score on this scale ranges from -36 to +36 and allows for different classes: non-apathetic (score -36 to -22); tendency to apathy (-21 to -17); moderate apathy (-16 to -10); and severe apathy (-9 to +36).
Improvement of the score at the Calgary Depression Scale for Schizophrenia (CDSS) at 1 month | Change between Baseline and 1 month
  The Calgary Depression Scale for Schizophrenia (CDSS, Addington et al., 1993; validated in French; Bernard et al., 1998) is a nine-item structured interview assessing depression in schizophrenia that measures the severity of symptoms such as depressed mood, hopelessness, guilt, insomnia and suicide.
Improvement of the score at the Calgary Depression Scale for Schizophrenia (CDSS) at 3 months | Change between Baseline and 3 months
  The Calgary Depression Scale for Schizophrenia (CDSS, Addington et al., 1993; validated in French; Bernard et al., 1998) is a nine-item structured interview assessing depression in schizophrenia that measures the severity of symptoms such as depressed mood, hopelessness, guilt, insomnia and suicide.
Improvement of the score at the Calgary Depression Scale for Schizophrenia (CDSS) at 6 months | Change between Baseline and 6 months
  The Calgary Depression Scale for Schizophrenia (CDSS, Addington et al., 1993; validated in French; Bernard et al., 1998) is a nine-item structured interview assessing depression in schizophrenia that measures the severity of symptoms such as depressed mood, hopelessness, guilt, insomnia and suicide.
Improvement in the " negative symptoms " sub-score of the Positive And Negative Syndrome Scale (PANSS, Kay et al., 1987) at 1 month | Change between Baseline and 1 month
  The Positive And Negative Syndrome Scale is a scale hetero-evaluation of positive and negative symptomatology and general psychopathology in schizophrenia, consisting of 30 items, sides 1 to 7. The higher the score, the more severe the symptomatology. This scale provides scores on three syndromic dimensions: positive (7 items), negative (7 items) and positive (7 items), and general psychopathology (16 items) from a categorical and dimensional perspective.
Improvement in the " negative symptoms " sub-score of the Positive And Negative Syndrome Scale (PANSS, Kay et al., 1987) at 3 months | Change between Baseline and 3 months
  The Positive And Negative Syndrome Scale is a scale hetero-evaluation of positive and negative symptomatology and general psychopathology in schizophrenia, consisting of 30 items, sides 1 to 7. The higher the score, the more severe the symptomatology. This scale provides scores on three syndromic dimensions: positive (7 items), negative (7 items) and positive (7 items), and general psychopathology (16 items) from a categorical and dimensional perspective.
Improvement in the " negative symptoms " sub-score of the Positive And Negative Syndrome Scale (PANSS, Kay et al., 1987) at 6 months | Change between Baseline and 6 months
  The Positive And Negative Syndrome Scale is a scale hetero-evaluation of positive and negative symptomatology and general psychopathology in schizophrenia, consisting of 30 items, sides 1 to 7. The higher the score, the more severe the symptomatology. This scale provides scores on three syndromic dimensions: positive (7 items), negative (7 items) and positive (7 items), and general psychopathology (16 items) from a categorical and dimensional perspective.
increased percentage of personal goal attainment at 1 month | Change between Baseline and 1 month
  Participants will be asked to list the goals they wish to achieve in 6 months or less, and the percentage of goals achieved will be assessed by the question "Were you able to achieve your goals? "to determine whether or not each personal goal was achieved. The expected response is yes vs. no for each personal goal. This methodology corresponds to the one classically used in CM-II studies (Fritzsche et al., 2016).
increased percentage of personal goal attainment at 3 months | Change between Baseline and 3 months
  Participants will be asked to list the goals they wish to achieve in 6 months or less, and the percentage of goals achieved will be assessed by the question "Were you able to achieve your goals? "to determine whether or not each personal goal was achieved. The expected response is yes vs. no for each personal goal. This methodology corresponds to the one classically used in CM-II studies (Fritzsche et al., 2016).
increased percentage of personal goal attainment at 6 months | Change between Baseline and 6 months
  Participants will be asked to list the goals they wish to achieve in 6 months or less, and the percentage of goals achieved will be assessed by the question "Were you able to achieve your goals? "to determine whether or not each personal goal was achieved. The expected response is yes vs. no for each personal goal. This methodology corresponds to the one classically used in CM-II studies (Fritzsche et al., 2016).
Decreased perception of effort associated with achieving goals at 1 month | Change between Baseline and 1 month
  Participants will be asked to report on their perception of the effort associated with goal attainment as assessed by the question "Did achieving personal goals require you to make an effort? ". Responses will be on a 10-points Likert scale ranging from 1 ("no effort at all") to 10 ("a lot of effort").
Decreased perception of effort associated with achieving goals at 3 months | Change between Baseline and 3 months
  Participants will be asked to report on their perception of the effort associated with goal attainment as assessed by the question "Did achieving personal goals require you to make an effort? ". Responses will be on a 10-points Likert scale ranging from 1 ("no effort at all") to 10 ("a lot of effort").
Decreased perception of effort associated with achieving goals at 6 months | Change between Baseline and 6 months
  Participants will be asked to report on their perception of the effort associated with goal attainment as assessed by the question "Did achieving personal goals require you to make an effort? ". Responses will be on a 10-points Likert scale ranging from 1 ("no effort at all") to 10 ("a lot of effort").

CONTACTS AND LOCATIONS:
Locations (1):
- Montpellier University Hospital, Montpellier, France